CLINICAL TRIAL: NCT01843634
Title: A Pilot Study to Evaluate the Safety and Preliminary Evidence of a Therapeutic Effect of ODSH (2-0, 3-0, Desulfated Heparin) in Patients Receiving Induction or Consolidation Therapy for Acute Myeloid Leukemia
Brief Title: Ph I Safety and Efficacy of ODSH in Patients Receiving Induction or Consolidation Therapy for Acute Myeloid Leukemia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 63137
Record Dates: First submitted 2013-04-26; First posted 2013-04-30 (Estimated); Last update posted 2021-11-10 (Actual); Status verified 2015-08

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ODSH (Experimental)
  Interventions: Drug: ODSH

INTERVENTIONS:
Drug: ODSH

SUMMARY:
This is an open-label pilot study evaluating the safety and preliminary evidence of a therapeutic effect of ODSH (2-0, 3-0 desulfated heparin) in conjunction with standard induction and consolidation therapy for acute myeloid leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, previously untreated acute myeloid leukemia. Acute promyelocytic leukemia is excluded.
* No prior chemotherapy for acute myeloid leukemia; however, prior hydroxyurea to control white blood cell count is allowed.
* No prior chemotherapy or lenalinomide for treatment of myelodysplastic syndrome.
* Age: 18-70.
* ECOG Performance status 0-2
* Cardiac ejection fraction ≥ 50% (echocardiography or MUGA [multigated acquisition])
* Adequate hepatic and renal function (AST [aminotransferase], ALT [alanine aminotransferase], bilirubin and creatinine < 2.5 x upper normal limit).
* Able to provide informed consent and have signed an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* Patients with acute promyelocytic leukemia
* Patients with acute megakaryoblastic leukemia
* Patients with CNS (central nervous system) leukemia
* Presence of significant active infection or uncontrolled bleeding
* Any coexisting major illness or organ failure which contraindicates the dose-intensive chemotherapy regimen prescribed by this protocol
* Pre-existing liver disease that might impair ODSH clearance
* History of other active malignant disease within 5 years, other than cured basal cell carcinoma of the skin, cured in situ carcinoma of the cervix, or localized prostate cancer that has received definitive therapy. Such prostate cancer patients who are receiving hormonal therapy are eligible
* Use of recreational drugs or history of drug addiction, within the prior 6 months
* Known history of positive hepatitis B surface antigens or hepatitis C antibodies
* Known history of positive test for HIV (Human immunodeficiency virus) antibodies
* Psychiatric or neurologic conditions that could impair ability to give proper informed consent
* Presence of symptomatic congestive heart failure, unstable angina pectoris, symptomatic or poorly controlled cardiac arrhythmia
* Presence of uncontrolled thrombotic or hemorrhagic disorder
* A medical condition that requires the need to be on chronic anticoagulation
* Presence of any other serious uncontrolled medical disorder
* Treatment with any other investigational agent, or participation in another clinical trial within 28 days prior to study entry
* Pregnant or breast-feeding patients
* Patient with childbearing potential not using adequate contraception
* Hemorrhage risk that requires maintenance of platelet counts at 50,000/uL or higher.
* Any significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Safety by incidence of serious events | 12 months
Efficacy by time to platelet recovery | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Shami, M.D., Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States